CLINICAL TRIAL: NCT02712775
Title: Minocycline Administration During Human Liver Transplantation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study logistics
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCL-001
Record Dates: First submitted 2016-03-14; First posted 2016-03-18 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2016-03

CONDITIONS: Liver Disease
MeSH Terms: conditions — Liver Diseases | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Minocycline (Experimental): Experimental group will receive an infusion of minocycline, the investigational drug, through a needle in a vein in the arm at the dose of 200 mg at 1 h prior to transplantation and 100 mg 12 h and 24 h after transplantation. In addition, the donated liver will be flushed with 200 mg minocycline 1 h prior to transplantation.
  Interventions: Drug: Minocycline (yes/no)
- Saline (Placebo Comparator): Placebo group will receive an infusion of saline, a placebo, through a needle in a vein in the arm according to the same schedule. In addition, the donated liver will be flushed with saline 1 h prior to transplantation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minocycline (yes/no)
  Arms: Minocycline
Drug: Placebo — Saline
  Arms: Saline

SUMMARY:
Liver transplantation is the sole therapy for end-stage liver diseases and acute liver failure in children and adults. However, use of this life-saving technique is limited due to a severe shortage of donor livers. The number of transplants currently performed is approximately one-third of the number needed to accommodate the more than 16,000 patients awaiting an organ in the US. Over 20% of patients on the liver transplant waiting list die prior to transplantation due to organ shortages. The median waiting time in 2011 was over 300 days. Poor immediate graft function and primary non function (PNF) are clinically significant events, especially in recipients of marginal livers (elderly donors, extended cold storage time, or steatosis). PNF has dramatic effects on patient morbidity and mortality, necessitating prolonged and expensive stays in intensive care units, and re-transplantation is the only life-saving therapy in patients with failing liver grafts due to PNF. This further exerts greater burden on the already scarce donor organ pool. Furthermore, biliary strictures and ischemic cholangiopathy, as a result of severe ischemia reperfusion injury, cause prolonged hospital stay, long-term complications, and increased costs. Targeted treatments, such as the one proposed in this application, will reduce the need for re-transplantation, reduce biliary injury, and potentially increase the number of donor organs available.

DETAILED DESCRIPTION:
Liver transplantation is the sole therapy for end-stage liver diseases in children and adults. However, use of this life-saving technique is limited due to a severe shortage of donor livers and, consequently, over 1500 patients/year on waiting lists die prior to transplantation due to organ shortages. Also, poor immediate graft function remains a persistent problem especially in recipients of marginal livers, and biliary strictures evolving from reperfusion injury cause prolonged hospital stay, increased health care costs, and increased mortality. Furthermore, hepatic cold storage and reperfusion in transplantation settings cause mitochondrial dysfunction in liver cells, which constitutes a great risk for primary nonfunction and initial poor function after liver transplantation. The tetracycline derivative minocycline is a safe and widely used antibiotic that possesses cytoprotective effects through prevention of mitochondrial dysfunction in a variety of disease models. Recently, we showed that minocycline also protects against graft dysfunction and failure after orthotopic rat liver transplantation and against cell death after ischemia-reperfusion to cultured rat hepatocytes. Minocycline treatment specifically prevented mitochondrial dysfunction and increased graft and animal survival by blocking necrotic and apoptotic death pathways. Clinical studies indicating severe deterioration of mitochondrial function in livers during preservation provide a strong impetus to investigate minocycline as an effective agent to decrease injury and improve graft function after human clinical transplantation.

ELIGIBILITY:
Inclusion Criteria:

* All adult primary transplant recipients of solitary orthotopic liver transplants are considered for this study

Exclusion Criteria:

* Pediatric patients, fulminant hepatic failures, split livers, living donor liver transplants, multiple organs, known tetracycline hypersensitivity, and re-transplant patients are excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
AST | 6 month
  AST is the primary endpoint our study is powered to detect. Peak AST >1500 IU/L is associated with clinical sequel of IRI such as severe graft dysfunction and complications.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Chavin, MD, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States